CLINICAL TRIAL: NCT01479569
Title: Real-time MRI Pericardiocentesis Using Passive Needles
Brief Title: Pericardiocentesis With Magnetic Resonance Imaging
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120025; 12-H-0025
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2017-02-17

CONDITIONS: Cardiac Magnetic Resonance Imaging
Keywords: MRI Catheterization; Pericardiocentesis; MRI Safety; Cardiac Magnetic Resonance Imaging
MeSH Terms: interventions — Pericardiocentesis

INTERVENTIONS:
Procedure: Pericardiocentesis

SUMMARY:
Background:

- Pericardiocentesis uses a needle and small tube to drain fluid from space around the heart. The most common reason to perform this procedure is that the fluid is interfering with heart function. This procedure is usually guided by X-rays. However, researchers want to try the procedure using magnetic resonance imaging (MRI) instead of X-rays. MRI guidance may be more precise than X-rays, which can make the procedure easier and more effective.

Objectives:

- To test whether MRI guidance can improve pericardiocentesis.

Eligibility:

- Individuals at least 18 years of age who need to have pericardiocentesis.

Design:

* Participants will have a physical exam before the procedure. Blood samples will be taken.
* The pericardiocentesis will be performed using MRI guidance. The procedure may take up to 2 hours.
* If for some reason the MRI guidance is not successful, participants will have the regular X-ray procedure. The MRI system will be used to take high-quality pictures afterward to check the results....

DETAILED DESCRIPTION:
Pericardiocentesis is a minimally invasive procedure to drain fluid from the pericardial space, created by the pericardial sac which cradles the heart. The most common reason to perform this procedure is that pericardial fluid is interfering with heart function. The next most common reason is to obtain pericardial fluid for testing to make a clinical diagnosis. Pericardiocentesis is performed using a long needle that may be guided by various means including blindly without imaging guidance, using electrocardiography electrodes to determine when the needle accidentally touches the heart, using echocardiography, using X-ray with- or without- contrast injections, or using a combination. Each has its advantages and limitations.

We have developed real-time magnetic resonance imaging (MRI) to guide heart catheterization with tissue visualization but without X-ray radiation. When used to guide needle access to the pericardial space or from there even into heart cavities, MRI provides superb imaging guidance. What is especially valuable about MRI is that it provides the entire thoracic context of needle access, allowing the operator to avoid critical structures including the liver, lung, pleural space, and heart muscle.

We have developed real-time magnetic resonance imaging (MRI) to guide heart catheterization in patients with tissue visualization but without X-ray radiation. We also have used these developments to guide needle access to the heart and pericardium in animal models.

In this protocol we test the safety and feasibility of pericardiocentesis in adult patients, using commercially available MRI-compatible (passive) needles.

If successful, this will enable more advanced minimally invasive procedures in adults and children.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult patients, age greater than or equal to 18
* Undergoing medically necessary diagnostic or therapeutic pericardiocentesis

EXCLUSION CRITERIA:

* Cardiogenic shock (sustained systolic blood pressure less than or equal to 80 mm Hg despite volume repletion on physical examination or requiring catecholamine support)
* Women who are pregnant or nursing
* Unable to undergo magnetic resonance imaging

  * Cardiac pacemaker or implantable defibrillator
  * Cerebral aneurysm clip
  * Neural stimulator (e.g. TENS-Unit)
  * Any type of ear implant
  * Ocular foreign body (e.g. metal shavings)
  * Metal shrapnel or bullet.
  * Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe for MRI

EXCLUSION CRITERIA FOR GADOLINIUM-BASED CONTRAST AGENTS:

* Renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73M(2) body surface area according to the Modification of Diet in Renal Disease criteria
* Glomerular filtration rate will be estimated using the MDRD 2005 revised study formula:

  --eGFR (mL/min/1.73M(2))=175x(standardized s(cr)) (-1.154) x (age) (-0.203) x 0.742 (if the subject is female) or x1.212 (if the subject is black)
* Subjects meeting this exclusion criterion may still be included in the study but may not be exposed to gadolinium-based contrast agents.

RATIONALE FOR SELECTION CRITERIA:

* This is a technical development study with the prospect of direct benefit to individual research subjects. The selection criteria are designed to minimize risk while attaining the scientific objectives of the study.
* Adult subjects are sought from among patients already undergoing medically necessary pericardiocentesis. Children are excluded from this first proof-of-concept experience to maximize safety; we anticipate a follow-on protocol that includes children.
* Subjects are excluded if they are not suitable for rapid entry into an interventional MRI environment, so mechanical ventilation and cardiogenic shock are exclusion criteria in this early experience.
* Subjects with renal excretory dysfunction might be injured by gadolinium exposure and are not exposed to gadolinium-based contrast agents. Pregnant subjects are excluded because of unknown risk and no benefit to a fetus. Magnetic resonance imaging will be used to guide pericardiocentesis, so subjects must be eligible to undergo magnetic resonance imaging safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11-08; Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
Reduce the pericardial effusion.

SECONDARY OUTCOMES:
To test the feasibility of navigating passive needles percutaneously into the periocardial space using real-time MRI and MRI-compatible needles.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Saikus CE, Lederman RJ. Interventional cardiovascular magnetic resonance imaging: a new opportunity for image-guided interventions. JACC Cardiovasc Imaging. 2009 Nov;2(11):1321-31. doi: 10.1016/j.jcmg.2009.09.002. PMID 19909937
- [Background] Ratnayaka K, Faranesh AZ, Guttman MA, Kocaturk O, Saikus CE, Lederman RJ. Interventional cardiovascular magnetic resonance: still tantalizing. J Cardiovasc Magn Reson. 2008 Dec 29;10(1):62. doi: 10.1186/1532-429X-10-62. PMID 19114017
- [Background] Guttman MA, Lederman RJ, Sorger JM, McVeigh ER. Real-time volume rendered MRI for interventional guidance. J Cardiovasc Magn Reson. 2002;4(4):431-42. doi: 10.1081/jcmr-120016382. PMID 12549231